CLINICAL TRIAL: NCT00574990
Title: Minimizing Harm From ADEs by Improving Nurse-Physician Communication
Acronym: MED-COMM
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: NRI 05-275
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Interdisciplinary Communication; Management, Medication Therapy
Keywords: Interdisciplinary Communication; Safety Management; Management, Medication Therapy; Cooperative Behavior; Drug Therapy Management; Physician Nurse Relationships; Side Effects; Hospital Information Systems; Documentation; Quality Assurance, Health Care
MeSH Terms: conditions — Cooperative Behavior

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- VA Physicians: VA providers who had worked at least one year in the VA and were familiar with the VA's electronic health record, CPRS.
- VA Nurses: VA nurses who had worked at least one year in the VA and were familiar with the VA's electronic health record, CPRS.
- VA Pharmacists: VA pharmacists who had worked at least one year in the VA and were familiar with the VA's electronic health record, CPRS.

SUMMARY:
The purpose of this research study is to examine the clinical processes of care involved with the sharing and communicating of medication management information in the inpatient setting between nurses, pharmacists and physicians. The study is unique in that few studies have examined communication content and processes in depth and in relation to specific clinical care. The study will be conducted in two phases. The first phase involves using three focus groups across three sites (a total of nine) each involving between 6-8 individuals to examine perceptions regarding role and procedures associated with medication management. The focus group discussions will be tape-recorded and analyzed using qualitative methods. The information gleaned will assist us in identifying patterns of problems in enhancing the sharing of information, to develop better measures for assessing communication as well as designing effective interventions to enhance communication.

In the second phase of the study, 400 2-4 hour time slots will be randomly selected over about a 5-week period for nursing staff and 500 events over a 6-week period for physicians to conduct ethnographic observations during which specific communication events will be recorded and coded. Every effort will be made to minimize interruptions during clinical care. This research has not been done in terms of medication management content in the inpatient setting (non-ICU).

DETAILED DESCRIPTION:
Background:

Medication management is a complex clinical task. It requires substantial collaboration and coordination between physicians, nurses and pharmacists. Addressing ineffective communication has been identified by the Institute of Medicine as a high priority. Ineffective communication regarding medication management coordination can result in increased medication errors, rates of adverse drug events (ADEs), delays in treating adverse drug events and less effective treatment. ADEs are frequent in hospitalized patients, ranging from less than 3% to over 32%. The purpose of this study was to evaluate communication patterns associated with medication management between providers, physicians and pharmacists in the inpatient setting.

Objectives:

Specific Aim 1. Assess clinicians' beliefs and concerns regarding the role of communication in preventing, detecting and managing ADEs in elderly inpatients (focus groups).

Specific Aim 2. Evaluate and characterize communication events between VA nurses, physicians and pharmacists in an inpatient medicine setting (ethnographic observation).

Methods:

Phase 1: Focus Groups Design: The design of this study was qualitative and used focus group methodology.

Settings: Three VA sites that differed in size, location and academic affiliation were selected.

Participants: Three focus groups were conducted at each site (one each of pharmacists, nurses and physicians). A total of 19 nurses, 16 pharmacists and 13 doctors participated.

Phase 2: Observation Design: The design of this study was quantitative and descriptive. Settings: Two inpatient units at the VA Salt Lake City Health Care System (medicine and telemetry).

Participants: Twelve residents were selected randomly from each of the 4 medical teams, 19 nurses were selected randomly from the two in-patient medicine wards, and 8 clinical pharmacists (the total number of clinical pharmacists available) agreed to participate.

Status:

All data have been collected and initial analyses has been completed.

ELIGIBILITY:
Inclusion Criteria:

Providers who are working in the VA on the inpatient setting, including pharmacists, nurses, and physicians.

Exclusion Criteria:

Staff who have worked at the VA less than 1 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: VA Physicians, Nurses, and Pharmacists had worked at least one year in the VA and were familiar with the VA's electronic health record, CPRS.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlene R Weir, PhD RN, Principal Investigator — Salt Lake City
Locations (3):
- United States (3):
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Medical Center, Asheville, Asheville, North Carolina
  - Salt Lake City, Salt Lake City, Utah

REFERENCES:
- [Result] Flaherty JH, Shay K, Weir C, Kamholz B, Boockvar KS, Shaughnessy M, Shapiro R, Gordon S, Stein J, Rudolph JL; VA Delirium Working Group. The development of a mental status vital sign for use across the spectrum of care. J Am Med Dir Assoc. 2009 Jul;10(6):379-80. doi: 10.1016/j.jamda.2009.04.001. No abstract available. PMID 19560714
- [Result] Vogelsmeier A, Pepper GA, Oderda L, Weir C. Medication reconciliation: A qualitative analysis of clinicians' perceptions. Res Social Adm Pharm. 2013 Jul-Aug;9(4):419-30. doi: 10.1016/j.sapharm.2012.08.002. Epub 2012 Oct 23. PMID 23089295

RESULTS

PARTICIPANT FLOW:
Groups:
- VA Physicians: VA Physicians who have spent at least one year in the VA and be familiar with the VA's electronic health record, CPRS.
Period: Overall Study
Arm/Group | VA Physicians | VA Nurses | VA Pharmacists
Started | 12 | 19 | 8
Completed | 12 | 19 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VA Physicians: VA physicians who had worked at least one year in the VA and were familiar with the VA's electronic health record, CPRS.
- Total: Total of all reporting groups
Arm/Group | VA Physicians | VA Nurses | VA Pharmacists | Total
Number analyzed (Participants) | 12 | 19 | 8 | 39
Age, Customized [Number; unit: participants]
  18 to 75 years | 12 | 19 | 8 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — No demographics were collected including gender. | NA — No demographics were collected including gender. | NA — No demographics were collected including gender. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — No demographics were collected including gender. | NA — No demographics were collected including gender. | NA — No demographics were collected including gender. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 19 | 8 | 39

OUTCOME MEASURES:

1. Primary Outcome: Incident Rate for Communication Events
Description: Observation periods were approximately two-hours long. Some providers were observed more than once. The number of communication events were counted per each observation period.
Time Frame: 6 months
Population: Participants were providers who had worked at least one year in the VA and were familiar with the VA's electronic health record, CPRS.
Measure: Mean (Standard Deviation); unit: mean events per observation
Groups:
- Physicians; Nurses; Pharmacists: Participants were providers who had worked at least one year in the VA and were familiar with the VA's electronic health record, CPRS.
Arm/Group | Physicians | Nurses | Pharmacists
Number analyzed (Participants) | 12 | 19 | 8
mean events per observation | 47.6 (21.26) | 34.74 (9.93) | 34.07 (12.88)
Statistical Analysis 1: Comparison: Physicians vs Nurses vs Pharmacists; Descriptive counts and chi squared were done on the observation data; Test type: Superiority or Other; p = 0.01, Chi-squared — Differences between roles and communication event content were assessed by Chi squared; chi square = 12.99, Standard Error of Mean 1.4

2. Secondary Outcome: Overall Involvement in Conversation by Roles
Description: The number of communication events was recorded on electronic notepads during each observation period. The communication events recorded included: a) physicians to physicians, to nurses, to pharmacists, and to patients; b) nurses to nurses, to physicians, to pharmacists, and to patients; and c) pharmacists to pharmacists, to physicians, to nurses, and to patients. The percentage of each of these types of verbal communications was calculated from the total number of communication events.
Time Frame: 6 months
Measure: Number; unit: percentage of role involvement in event
Arm/Group | VA Physicians | VA Nurses | VA Pharmacists
Number analyzed (Participants) | 12 | 19 | 8
percentage of role involvement in event
  VA Physicians | 31 | 21 | 58
  VA Nurses | 12 | 23 | 9
  VA Pharmacists | 20 | 6 | 12
  VA Inpatient Patients | 6 | 27 | 8

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- VA Physicians: VA Physicians who had worked at the VA for at least one year and were familiar with the VA's electronic health record, CPRS.
- VA Nurses: VA Nurses who had worked at the VA for at least one year and were familiar with the VA's electronic health record, CPRS.
- VA Pharmacists: VA Pharmacists who had worked at the VA for at least one year and were familiar with the VA's electronic health record, CPRS.
Arm/Group | VA Physicians | VA Nurses | VA Pharmacists
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/19 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/19 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes